CLINICAL TRIAL: NCT04244188
Title: Simulation of Stent-graft Deployment in Aortic Arch Aneurysms
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN032019/CHUSTE
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Aortic Arch Aneurysm
Keywords: Numerical simulation; stent-graft; aortic arch aneurysms
MeSH Terms: conditions — Aneurysm, Aortic Arch

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated for aortic arch aneurysms: Patients treated for aortic arch aneurysms by double branched endovascular repair (Bolton Medical) will be included.
  Interventions: Other: Collection of datas

INTERVENTIONS:
Other: Collection of datas — Collection of datas: pre- and postoperative scanner and endoprosthesis characteristics

SUMMARY:
Total endovascular repair of the aortic arch represents a promising option for patients ineligible to open surgery. Custom-made design of stent-grafts (SG), such as the Terumo Aortic® RelayBranch device (DB), requires complex preoperative measures. Accurate SG deployment is required to avoid intraoperative or postoperative complications, which is extremely challenging in the aortic arch. In that context, the investigators aim is to develop a computational tool able to predict SG deployment in such highly complex situations. Four patient-specific cases will be performed with complete deployment of the DB and its bridging stents in aneurysmal aortic arch. Deviations of simulation predictions from actual stent positions will be estimated based on post-operative scan and a sensitivity analysis will be performed to assess the effects of material parameters. If good agreement between simulation and reality is obtained, numerical simulations will show their ability to successfully predict the DB deployment in complex anatomy. The results will emphasize the potential of computational simulations to assist practitioners in planning and performing complex and secure interventions.

DETAILED DESCRIPTION:
The process of numerical simulation of double-branched device in aortic arch aneurysm involves: (i) aortic arch segmentation with data from the preoperative CT-scan (ii) numerical modeling of the actual stentgraft used to treat the patient (iii) simulation of stentgraft deployment in aortic arch (iv) validation of simulation results based on post-operative CT scan images The goal of this study is to develop a numerical model of stentgraft deployment able to predict the actual deployement of the double branched device in aortic arch aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* Aortic arch aneurysms suitable for treatment using double-branched device Bolton

Exclusion Criteria:

* Failure to generate an adequate FE model of patient arteries (no preoperative multidetector contrast-enhanced CT-scan available, preoperative CT-scan slice thickness greater than 1mm, preoperative CT- scan with artifacts)
* dissected aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for aortic arch aneurysms by double branched endovascular repair (Bolton Medical) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
In vitro versus stimulation test | Day 0
  To compare Vascutek in vitro validation test to the simulation of this test, the proportion of fLenestrations where |L3 - L2| and |C3 - C2| are less or equal to 2.5mm will be analysed.
  L3=distal edge of celiac trunk (L) after first simulation, stent-graft deployment in rigid aorta L2=distal edge of celiac trunk (L) after final custom stent-graft design, after in vitro tests

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Noël ALBERTINI, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- CHU Saint-Etienne, Saint-Etienne, France
- Rinjstate Hopital, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Derycke L, Perrin D, Cochennec F, Albertini JN, Avril S. Predictive Numerical Simulations of Double Branch Stent-Graft Deployment in an Aortic Arch Aneurysm. Ann Biomed Eng. 2019 Apr;47(4):1051-1062. doi: 10.1007/s10439-019-02215-2. Epub 2019 Jan 31. PMID 30706308